CLINICAL TRIAL: NCT02561481
Title: Sulforaphane Treatment of Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Andrew Zimmerman, Clinical Professor of Pediatrics and Neurology, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H00007832; AR140087 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulforaphane (Active Comparator): Sulforaphane (SF) will be administered once a day orally in an approximate dose of 1 µmol/lb (2.2 kg µmol/kg) body weight. Each SF tablet will contain 125 mg broccoli seed powder (equivalent to ~ 15 µmol SF). The total dose per day will depend on participants' body weight:
  30-50 lb: 3 tablets (45 µmol/day) 50-70 lb: 4 tablets (60 µmol/day) 70-90 lb: 6 tablets (90 µmol/day) 90-110 lb: 7 tablets (105 µmol/day) 110-130 lb: 8 tablets (120 µmol/day)
  For pilot study, all participants (n=10) will receive SF for 14 days. For main clinical trial, 25 participants will randomly receive SF for 15 weeks (phase 1). During phase 2, a single-arm crossover from placebo to sulforaphane arm will take place, and all participants will receive SF from 15-30 weeks.
  Interventions: Drug: Sulforaphane
- Placebo (Placebo Comparator): Placebo tablets identical in size and similar in appearance to the active tablets will be used. Number of placebo tablets will be equivalent to the active tablets depending on participants' body weight.
  For the main clinical trial, 25 participants will be randomly allocated to receive placebo for 15 weeks (phase 1). During phase 2, a single-arm crossover from placebo arm to sulforaphane arm will take place, and all participants will receive sulforaphane from 15-30 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulforaphane — See under active arm description
  Arms: Sulforaphane
Drug: Placebo — See under placebo arm description
  Arms: Placebo

SUMMARY:
ASD is a diverse disorder starting in early childhood and characterized by social communication impairment as well as restricted interests and repetitive behaviors. It affects 1:68 children and is an enormous medical and economic problem for which there is no established, mechanism-based treatment. Sulforaphane is an isothiocyanate derived from broccoli, and has potent activity in transcriptionally up-regulating genes that control mechanisms whereby aerobic cells protect themselves against oxidative stress, mitochondrial dysfunction, and inflammation.

This study is a clinical trial of oral sulforaphane (as broccoli seed powder) in 50 boys and girls (3-12 years) with ASD in 3 phases over 36 weeks. In Phase 1, 25 children will receive active drug and 25 will receive placebo for 15 weeks; in Phase 2, all children will receive sulforaphane from 15-30 weeks; in Phase 3, children will receive no treatment for 6 weeks. Study visits will take place at screening, 7, 15, 22, 30 and 36 weeks, when the Ohio Autism Clinical Clinical Impressions Scale - Severity and Improvement (OACIS-S and OACIS-I), Aberrant Behavior Checklist (ABC) and Social Responsiveness Scale (SRS) will be recorded. Children will be monitored with physical examinations and for toxicity with clinical laboratory studies and examine possible biomarkers: Nuclear factor-erythroid factor 2 (Nrf2), oxidative stress and mitochondrial function, the mechanistic target of rapamycin (mTOR) pathway and cytokine expression. In addition, prior to the main clinical trial, a pilot study will be carried out in 10 children with ASD, 6-12 years of age, who will receive sulforaphane, 2.2 micromoles/kg daily for 14 days. Blood and urine samples before and at the end of treatment will be collected, in order to measure several parameters that are likely to demonstrate expected effects of sulforaphane, to standardize the assays and procedures, and to determine the most effective measures.

DETAILED DESCRIPTION:
Background: ASD is a diverse disorder starting in early childhood and characterized by social communication impairment as well as restricted interests and repetitive behaviors. It affects 1:68 children and is an enormous medical and economic problem for which there is no established, mechanism-based treatment. Sulforaphane is an isothiocyanate derived from broccoli, and has potent activity in transcriptionally up-regulating genes that control mechanisms whereby aerobic cells protect themselves against oxidative stress, mitochondrial dysfunction, and inflammation.

Hypothesis: Based on the observation that fever is frequently associated with behavioral improvements in children with ASD, it is hypothesized that sulforaphane might lead to functional improvements in ASD because it can up-regulate cell-protective responses, such as heat shock proteins and related mechanisms that are also up-regulated during fever. These mechanisms are central to multiple cellular processes in the central nervous system, including synaptic transmission, and may improve long-range cerebral cortical connectivity, which is depressed in ASD.

Specific aims: The 3 specific aims in this study are: 1) To determine if there are measurable effects on social responsiveness and problem behaviors during treatment of children with sulforaphane; 2) To determine if treatment with sulforaphane in children is safe and well tolerated; and 3) To elucidate cellular biomarkers that respond to treatment with sulforaphane.

Design: This is a randomized, double blind, single-arm crossover phase 1/2 clinical trial of orally administered sulforaphane (as broccoli seed powder) in 50 boys and girls (3-12 years) with ASD in 3 phases over 36 weeks.

In Phase 1, 25 children will receive active drug and 25 will receive placebo for 15 weeks; in Phase 2, all children will receive sulforaphane from 15-30 weeks; in Phase 3, children will receive no treatment for 6 weeks. Study visits will take place at screening, 7, 15, 22, 30 and 36 weeks, when the Ohio Autism Clinical Clinical Impressions Scale - Severity and Improvement (OACIS-S and OACIS-I), Aberrant Behavior Checklist (ABC) and Social Responsiveness Scale (SRS) will be recorded.

The children will be monitored with physical examinations and for toxicity with clinical laboratory studies and examine possible biomarkers: Nrf2, oxidative stress and mitochondrial function, mTOR pathway and cytokine expression.

In addition, prior to the main clinical trial, a pilot study will be performed in 10 children with ASD, 6-12 years of age, who will receive sulforaphane, 2.2 micromoles/kg daily for 14 days. Blood and urine samples before and at the end of treatment will be collected, in order to measure several parameters that are likely to demonstrate expected effects of sulforaphane, to standardize the assays and procedures, and to determine the most effective measures.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD) diagnosis of moderate or greater severity
* Age 3 through 12 years inclusive

Exclusion Criteria:

* Absence of a parent or legal guardian and consent
* Inability to speak/understand English language
* Seizure within 1 year of screening: This exclusion is based on the theoretical concern that cellular activation by sulforaphane might exacerbate seizures in patients with known seizure disorders. As noted in our previous trial of sulforaphane in young adult males, a seizure occurred in each of 2 participants: one during treatment (in a participant with a previously undisclosed seizure), the other 3 weeks after discontinuing sulforaphane.
* Impaired renal function (serum creatinine > 1.2 mg/dl), impaired hepatic function (SGOT/SGPT> 2x upper limit of normal), impaired thyroid function (Thyroid Stimulating Hormone (TSH) outside normal limits): This exclusion is based on a theoretical possibility of activation of underlying cellular metabolic abnormalities by sulforaphane. Current infection or treatment with antibiotics: this exclusion is to avoid complications of inter-current illness that may occur due to the clinical trial or obscure possible effects of sulforaphane.
* Medications that may modify the course or testing of ASD parameters (e.g., prednisone): This exclusion is necessary in order not to interfere with or complicate effects of sulforaphane.
* Chronic medical disorder (e.g., cardiovascular disease, stroke or diabetes) or major surgery within 3 months prior to enrollment: Serious medical illness in the child may be complicated by the clinical trial and make it difficult to discern a change in ASD associated with treatment.
* Less than 3 years or more than 13 years of age: this age range was selected to cover the ages from usual diagnosis of ASD up to adolescence.
* A diagnosis of autism spectrum disorder of mild severity (for example, earlier categories of Asperger disorder, Pervasive Developmental Disorder - Not Otherwise Specified (PDD-NOS)), according to Autism Diagnostic Observation Schedule (ADOS) criteria.
* Prisoners
* Pregnant women

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Zimmerman, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065
- [Result] Liu H, Zimmerman AW, Singh K, Connors SL, Diggins E, Stephenson KK, Dinkova-Kostova AT, Fahey JW. Biomarker Exploration in Human Peripheral Blood Mononuclear Cells for Monitoring Sulforaphane Treatment Responses in Autism Spectrum Disorder. Sci Rep. 2020 Apr 2;10(1):5822. doi: 10.1038/s41598-020-62714-4. PMID 32242086
- [Derived] Zimmerman AW, Singh K, Connors SL, Liu H, Panjwani AA, Lee LC, Diggins E, Foley A, Melnyk S, Singh IN, James SJ, Frye RE, Fahey JW. Randomized controlled trial of sulforaphane and metabolite discovery in children with Autism Spectrum Disorder. Mol Autism. 2021 May 25;12(1):38. doi: 10.1186/s13229-021-00447-5. PMID 34034808

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulforaphane: Sulforaphane (SF) will be administered once a day orally in an approximate dose of 1 µmol/lb (2.2 kg µmol/kg) body weight. Each SF tablet will contain 125 mg broccoli seed powder (equivalent to ~ 15 µmol SF). The total dose per day will depend on participants' body weight:
  30-50 lb: 3 tablets (45 µmol/day) 50-70 lb: 4 tablets (60 µmol/day) 70-90 lb: 6 tablets (90 µmol/day) 90-110 lb: 7 tablets (105 µmol/day) 110-130 lb: 8 tablets (120 µmol/day)
  For pilot study, all participants (n=10) will receive SF for 14 days. For main clinical trial, 25 participants will randomly receive SF for 15 weeks (phase 1). During phase 2, a single-arm crossover from placebo to sulforaphane arm will take place, and all participants will receive SF from 15-30 weeks.
  Sulforaphane: See under active arm description
- Placebo: Placebo tablets identical in size and similar in appearance to the active tablets will be used. Number of placebo tablets will be equivalent to the active tablets depending on participants' body weight.
  For the main clinical trial, 25 participants will be randomly allocated to receive placebo for 15 weeks (phase 1). During phase 2, a single-arm crossover from placebo arm to sulforaphane arm will take place, and all participants will receive sulforaphane from 15-30 weeks.
  Placebo: See under placebo arm description
Period: Pilot Trial
Arm/Group | Sulforaphane | Placebo
Started (Pilot study) | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0
Period: Main Trial - Double Blind Phase
Arm/Group | Sulforaphane | Placebo
Started | 25 | 25
Completed | 22 | 23
Not Completed | 3 | 2
Period: Main Trial - Open Label Phase
Arm/Group | Sulforaphane | Placebo
Started | 45 | 0
Completed | 32 | 0
Not Completed | 13 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane | Placebo | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (3.0) | 7.0 (2.5) | 7.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 15 | 32
  Other (asian, mixed, and unknown) | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Ohio Autism Clinical Impressions Scale - Improvement (OACIS-I) Average Score From Baseline
Description: The Ohio Autism Clinical Impressions Scale-Severity (OACIS-S) rates severity of symptoms in 10 categories: general level of autism, social interaction, aberrant and repetitive behavior, verbal and nonverbal communication, hyperactivity, anxiety, sensory sensitivities and restricted and narrow interests. Each category is rated from 1 (normal) to 7 (most severe). The OACIS-S was a reference at follow up visits when the OACIS-Improvement was compared to the OACIS-S, from 1 to 7: 4 was no change; 3 to 1 minimal to marked improvement and 5 to 7 minimal to marked worsening. The numerical score of the OACIS-S is independent and unrelated quantitatively to the OACIS-I. For analysis, the OACIS-I general score and subscale values were recoded, in which 4 (no change) was recoded as 0; 3 to 1 were recoded as +1 to +3 to denote improvement, and 5 to 7 were recoded as -1 to -3 for worsening.
Time Frame: 7 weeks, 15 weeks, 22 weeks, 30 weeks, 36 weeks
Population: Patients started dropping out at subsequent visits so the number analyzed at latter visits is less
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale
  7 weeks | 0.28 (0.67) | 0.28 (0.57)
  15 weeks | 0.28 (0.57) | 0.33 (0.69)
  22 weeks: number analyzed (Participants) | 17 | 17
  22 weeks | 0.47 (0.72) | 0.59 (0.71)
  30 weeks: number analyzed (Participants) | 16 | 16
  30 weeks | 0.47 (0.67) | 0.69 (0.77)
  36 weeks: number analyzed (Participants) | 14 | 14
  36 weeks | 0.29 (0.73) | 0.29 (0.61)

2. Secondary Outcome: OACIS-I Response Rate on Aberrant Behaviors Subscale
Description: See above in the primary outcome measure for a description of OACIS-I scale. This section describes the change from baseline of the OACIS-I subdomain of aberrant behaviors. This subdomain has a range of 1 to 7 - 1 is extremely improved from baseline, 7 is extremely worse from baseline, and 4 is no change. For analysis, the OACIS-I general score and subscale values were recoded, in which 4 (no change) was recoded as 0; 3 to 1 were recoded as +1 to +3 to denote improvement, and 5 to 7 were recoded as -1 to -3 for worsening.
Time Frame: 7 weeks, 15 weeks, 22 weeks, 30 weeks, 36 weeks
Population: Patients started dropping out at subsequent visits so the number analyzed at latter visits is less
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale
  7 weeks | 0.06 (0.42) | 0.28 (0.57)
  15 weeks | 0.22 (0.43) | 0.33 (0.69)
  22 weeks: number analyzed (Participants) | 17 | 17
  22 weeks | 0.59 (0.80) | 0.53 (0.87)
  30 weeks: number analyzed (Participants) | 16 | 16
  30 weeks | 0.63 (0.89) | 0.59 (0.84)
  36 weeks: number analyzed (Participants) | 14 | 14
  36 weeks | 0.14 (0.77) | 0.14 (0.53)

3. Secondary Outcome: OACIS-I Response Rate on Social Communication Subscale
Description: See above in the primary outcome measure for a description of OACIS-I scale. This section describes the change from baseline of the OACIS-I subdomain of social communication. This subdomain has a range of 1 to 7 - 1 is extremely improved from baseline, 7 is extremely worse from baseline, and 4 is no change. For analysis, the OACIS-I general score and subscale values were recoded, in which 4 (no change) was recoded as 0; 3 to 1 were recoded as +1 to +3 to denote improvement, and 5 to 7 were recoded as -1 to -3 for worsening.
Time Frame: 7 weeks, 15 weeks, 22 weeks, 30 weeks, 36 weeks
Population: Patients started dropping out at subsequent visits so the number analyzed at latter visits is less
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale
  7 weeks | 0.33 (0.69) | 0.56 (0.70)
  15 weeks | 0.44 (0.70) | 0.56 (0.62)
  22 weeks: number analyzed (Participants) | 17 | 17
  22 weeks | 0.65 (0.79) | 1.35 (0.61)
  30 weeks: number analyzed (Participants) | 16 | 16
  30 weeks | 0.94 (0.83) | 1.25 (0.61)
  36 weeks: number analyzed (Participants) | 14 | 14
  36 weeks | 0.32 (0.61) | 0.61 (0.66)

4. Secondary Outcome: Change in Total Aberrant Behavior Checklist Score From Baseline
Description: Aberrant Behavior Checklist (ABC) is a 58 item scale that primarily evaluates how aberrant or abnormal a patient's daily behaviors are. The items evaluate behaviors as they pertain to irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech. Each item is scored on a scale of 0 to 3, with 0 being better outcome and 3 being worse outcome. The score from each item is added up to calculate a total score. This outcome describes change in total ABC score from baseline at each follow up visit. The scores from all items are added to calculate a total score (0 to 174). This outcome describes change in total ABC score from baseline at each follow up visit.
Time Frame: 7 weeks, 15 weeks, 22 weeks, 30 weeks, 36 weeks
Population: Patients started dropping out at subsequent visits so the number analyzed at later visits is less
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale
  7 weeks | -6 (3.4) | -16.23 (14.02)
  15 weeks: number analyzed (Participants) | 14 | 14
  15 weeks | -22.6 (10.34) | -11.68 (5.40)
  22 weeks: number analyzed (Participants) | 15 | 15
  22 weeks | -36.33 (14.55) | -22.4 (15.45)
  30 weeks: number analyzed (Participants) | 11 | 11
  30 weeks | -22.8 (13.5) | -10.29 (9.97)
  36 weeks: number analyzed (Participants) | 3 | 3
  36 weeks | 1.14 (3.53) | -7.8 (5.56)

5. Secondary Outcome: Change in Total SRS-2 Score From Baseline
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item scale that measures total scores as well as subscales: four social behaviors (awareness, cognition, communication and motivation) and autistic mannerisms. Each item is rated from 1 to 4 (not true to almost always true) on worksheets that are blinded to the rater with respect to values. Total and subscale scores are calculated as raw scores and can be converted to T-scores. Raw scores (range 0-180) are reported here (unadjusted for general population, since all children had ASD). Higher or lower values at follow up visits compared to baseline indicated worsening or improvement, respectively.
Time Frame: 7 weeks, 15 weeks, 22 weeks, 30 weeks, 36 weeks
Population: Patients dropped out (or families did not return forms) at subsequent visits so the number analyzed at later visits is less.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale
  7 weeks | 1.14 (5.33) | -8.06 (7.89)
  15 weeks: number analyzed (Participants) | 21 | 22
  15 weeks | -16.86 (10.56) | -7.92 (4.45)
  22 weeks: number analyzed (Participants) | 20 | 18
  22 weeks | -14.61 (9.90) | -13.67 (11.23)
  30 weeks: number analyzed (Participants) | 15 | 16
  30 weeks | -19.83 (15.0) | -18.59 (11.57)
  36 weeks: number analyzed (Participants) | 9 | 8
  36 weeks | 0.80 (3.30) | -19.59 (10.17)

6. Secondary Outcome: Dithiocarbamate Plasma Concentration Detected by Cyclocondensation at Each Visit
Description: Sulforaphane (and other isothiocyanates, ITC) are conjugated by glutathione (GSH) which then undergoes further enzymatic modifications to give rise sequentially to the cysteinylglycine-, cysteine- and N-acetylcysteine-ITC conjugates, all of which are dithiocarbamates (DTC) and are detected in the cyclocondensation reaction-HPLC assay.
Time Frame: Week 0, Week 7, Week 15, Week 22, Week 30, Week 36
Population: Number analyzed varied due to participants who dropped out, their blood samples could not be obtained, or data could not be obtained from the assay.
Measure: Mean (Standard Deviation); unit: nmol DTC (Dithiocarbamates)/ml
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 24
nmol DTC (Dithiocarbamates)/ml
  Week 0 | 0.007 (0.008) | 0.006 (0.008)
  Week 7: number analyzed (Participants) | 22 | 22
  Week 7 | 0.299 (0.297) | 0.003 (0.005)
  Week 15 | 0.329 (0.350) | 0.005 (0.008)
  Week 22: number analyzed (Participants) | 19 | 20
  Week 22 | 0.248 (0,232) | 0.205 (0.253)
  Week 30: number analyzed (Participants) | 22 | 20
  Week 30 | 0.165 (0.183) | 0.214 (0.228)
  Week 36: number analyzed (Participants) | 15 | 16
  Week 36 | 0.015 (0.024) | 0.008 (0.012)

7. Secondary Outcome: Comparison of Free Reduced Glutathione (GSH), Total GSH, Oxidized Glutathione (GSSG) at Week 0 and 15
Description: F-statistic calculated by comparison of Free Reduced GSH, Total GSH and oxidized Glutathione (GSSG) of Week 15 to Week 0.
Time Frame: Week 0 and Week 15
Measure: Number; unit: F-statistic
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
F-statistic
  Free Reduced GSH | 1.51 | 0.11
  Total GSH | 0.00 | 0.08
  GSSG | 1.97 | 0.46

8. Secondary Outcome: Free GSH:GSSG and Total GSH:GSSG Ratios at Week 15
Description: Ratios of free GSH:GSSG and total GSH:GSSG were calculated by obtaining ratios of f-statistic scores from baseline to week 15 between free reduced GSH and GSSG and between total GSH and GSSG.
Time Frame: Week 15
Measure: Number; unit: F-statistic
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
F-statistic
  Free GSH:GSSG | 12.72 | 0.87
  Total GSH:GSSG | 5.16 | 0.03

9. Other Pre Specified Outcome: NQO1: NAD(P)H:Quinone Oxidoreductase-1
Description: Cytoprotective enzyme regulated by nuclear factor erythroid 2-related factor 2 (Nrf2), the master regulator of cellular redox homeostasis and an inhibitor of a key pro-inflammatory pathway, of which both functions are critical factors in the neuropathology of ASD. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Groups:
- Sulforaphane: Children receiving sulforaphane 0 - 30 weeks
- Placebo: Children receiving placebo from 0 - 15 weeks; received sulforaphane (SF) from 16 - 30 weeks.
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0 (baseline): number analyzed (Participants) | 21 | 18
  Week 0 (baseline) | 2.23 (0.18) | 2.25 (0.22)
  Week 15: number analyzed (Participants) | 21 | 23
  Week 15 | 2.19 (0.16) | 2.14 (0.20)
  Week 30: number analyzed (Participants) | 19 | 23
  Week 30 | 2.15 (0.15) | 2.13 (0.11)

10. Other Pre Specified Outcome: xCT
Description: xCT (SLC7A11): Cystine/glutamate antiporter encoded by the SLC7A11 gene.Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Groups:
- Placebo: Children receiving placebo 0 - 15 weeks; sulforaphane from 16 - 30 weeks
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 17 | 23
  Week 0 | 0.24 (0.94) | 0.40 (0.71)
  Week 15: number analyzed (Participants) | 17 | 21
  Week 15 | 0.25 (0.65) | 0.30 (0.95)
  Week 30: number analyzed (Participants) | 18 | 21
  Week 30 | 0.24 (1.02) | 0.27 (1.00)

11. Other Pre Specified Outcome: HO-1 (Heme Oxygenase 1)
Description: HO-1 (heme oxygenase 1): an essential and Nrf2-dependent enzyme in heme catabolism. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 19 | 16
  Week 0 | 0.10 (1.21) | 0.27 (0.98)
  Week 15: number analyzed (Participants) | 20 | 20
  Week 15 | 0.74 (0.69) | 0.55 (0.48)
  Week 30: number analyzed (Participants) | 19 | 20
  Week 30 | 0.74 (0.56) | 0.30 (1.40)

12. Other Pre Specified Outcome: HSP70
Description: HSP70 (Heat shock protein 70) was examined because it is upregulated by SF in vitro. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 22 | 19
  Week 0 | 1.11 (0.29) | 0.99 (0.43)
  Week 15: number analyzed (Participants) | 21 | 23
  Week 15 | 1.33 (0.43) | 1.14 (0.30)
  Week 30: number analyzed (Participants) | 20 | 23
  Week 30 | 1.23 (0.34) | 1.20 (0.40)

13. Other Pre Specified Outcome: HSP27
Description: HSP27 (Heat shock protein 27) was examined because it is upregulated by SF in vitro. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30.
Population: N varies due to missing data, variable clinic visits or assay failure
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 13 | 11
  Week 0 | 0.21 (0.46) | -0.13 (0.98)
  Week 15: number analyzed (Participants) | 10 | 14
  Week 15 | 0.21 (0.63) | -0.83 (1.21)
  Week 30: number analyzed (Participants) | 8 | 10
  Week 30 | -0.47 (1.21) | -0.58 (1.46)

14. Other Pre Specified Outcome: IL-6
Description: IL-6 (interleukin 6) cytokine gene expression, a nuclear factor-kappa B - regulated inflammatory biomarker. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 22 | 19
  Week 0 | 1.76 (0.39) | 1.82 (0.30)
  Week 15: number analyzed (Participants) | 20 | 23
  Week 15 | 2.05 (0.28) | 1.87 (0.42)
  Week 30: number analyzed (Participants) | 20 | 23
  Week 30 | 1.99 (0.23) | 2.08 (0.22)

15. Other Pre Specified Outcome: IL-1β
Description: IL-1β: Interleukin-1 beta cytokine gene expression, a nuclear factor-kappa B - regulated inflammatory biomarker. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 22 | 17
  Week 0 | 0.90 (1.16) | 1.14 (1.11)
  Week 15: number analyzed (Participants) | 19 | 22
  Week 15 | 1.45 (0.59) | 1.47 (0.50)
  Week 30: number analyzed (Participants) | 15 | 21
  Week 30 | 1.50 (0.49) | 1.59 (0.43)

16. Other Pre Specified Outcome: Cox-2
Description: Cox-2 (cyclooxygenase-2): a nuclear factor-kappa B - regulated inflammatory biomarker. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure.
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 15 | 14
  Week 0 | 0.14 (0.86) | -0.20 (1.06)
  Week 15: number analyzed (Participants) | 9 | 16
  Week 15 | -0.07 (1.59) | 0.16 (0.66)
  Week 30: number analyzed (Participants) | 9 | 14
  Week 30 | -0.46 (1.57) | -0.17 (1.17)

17. Other Pre Specified Outcome: TNF-α
Description: TNF-α (Tumor necrosis factor alpha), a cytokine as inflammatory biomarker. Total cellular RNA was isolated from peripheral blood mononuclear cells (PBMCs) and complementary DNAs (cDNA) were synthesized. Quantitative real-time PCR analysis was performed using the Applied Biosystems QuantStudio™ 3 Real-Time PCR System (Thermo Fisher Scientiﬁc, Waltham, MA, USA). Relative mRNA expression was normalized to GAPDH. Gene expression was calculated using the comparative 2-ΔΔCT method.
Time Frame: Week 0, Week 15, Week 30
Population: N varies due to missing data, variable clinic visits or assay failure
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 22 | 23
log fold change
  Week 0: number analyzed (Participants) | 21 | 17
  Week 0 | 0.70 (1.00) | 0.91 (0.37)
  Week 15: number analyzed (Participants) | 21 | 22
  Week 15 | 0.98 (1.03) | 1.08 (0.49)
  Week 30: number analyzed (Participants) | 19 | 23
  Week 30 | 1.17 (0.79) | 1.10 (0.73)

ADVERSE EVENTS:
Time Frame: The pilot study took place over 2 weeks for each of 10 participants. The main study took place over 2 years, 6 months; 1/1/16 - 6/30/18 for 45 participants, each of whom was assessed from screening (time 0), 7, 15, 22 and up to 36 weeks for the final visit. Participants in the pilot study were followed for adverse events during regular clinical visits for at least 12 months after the study and none were reported.
Description: Adverse event reporting followed clinicaltrials.gov Definitions.
Arm/Group | Sulforaphane | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/23
Other Adverse Events (participants affected / at risk) | 8/32 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulforaphane (N=32) | Placebo (N=23)
Hashimoto thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) — Participant was found to have elevated TSH. He was withdrawn from the study and was taking placebos. He was treated and followed by a pediatric endocrinologist, who determined that this was unrelated to his participation in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulforaphane (N=32) | Placebo (N=23)
insomnia (Nervous system disorders) | 2 | NA — sleep disturbance
irritability (Nervous system disorders) | 2 | NA
taste/smell (General disorders) | 2 | NA — unable to tolerate taste/smell of tablets
gastrointestinal upset (Gastrointestinal disorders) | 2 | NA

LIMITATIONS AND CAVEATS:
The sample size was limited to 45 children with ASD and we could not impute missing data for those participants who were lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT02561481/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT02561481/ICF_001.pdf